CLINICAL TRIAL: NCT04964778
Title: A Comparison of Respiratory Status and Comfort of Various Patient Packaging and Transport Configurations on Horizontal Ground
Brief Title: SKED Physiology Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to secure funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00072899
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Comparison of Patient Packaging and Transport Methods
Keywords: SKED; transport configurations; comfort; respiratory status

STUDY DESIGN:
Intervention Model Description: Each subject will be packaged with SKED© only; SKED©+OSS-II©; SKED©+Vacuum mattress; SKED©+foam padding. Each arm will consist of the same interventions in a specified, but unique order. Each patient packaged within their respective systems as one unit will be subject to a 30 meter controlled drag over terrain chosen to mimic a standard dry backcountry extrication drag.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Arm1: SKED© only first (Experimental): Each participant will be packaged using a SKED© system with no assumed spinal injury. Each arm will consist of the same interventions in a specified, but unique order. Arm 1 will be in the following order: SKED© only; SKED©+OSS-II©; SKED©+Vacuum mattress; SKED©+foam padding
  Interventions: Device: SKED©
- Arm 2: SKED©+Vacuum mattress first (Experimental): Each participant will be packaged using a SKED© system with no assumed spinal injury. Each arm will consist of the same interventions in a specified, but unique order. Arm 2 will be in the following order: SKED©+Vacuum mattress; SKED©+OSS-II©; SKED©+foam padding, SKED© only
  Interventions: Device: SKED©
- Arm 3: SKED©+OSS-II© first (Experimental): Each participant will be packaged using a SKED© system with no assumed spinal injury. Each arm will consist of the same interventions in a specified, but unique order. Arm 3 will be in the following order: SKED©+OSS-II©;SKED©+Vacuum mattress; SKED© only; SKED©+foam padding
  Interventions: Device: SKED©
- Arm 4: SKED©+foam padding first (Experimental): Each participant will be packaged using a SKED© system with no assumed spinal injury. Each arm will consist of the same interventions in a specified, but unique order. Arm 4 will be in the following order: SKED©+foam padding, SKED©+Vacuum mattress; SKED© only; SKED©+OSS-II
  Interventions: Device: SKED©

INTERVENTIONS:
Device: SKED© — A SKED device is lightweight plastic stretcher used for moving patients through difficult terrain.

SUMMARY:
A SKED© is a stretcher typically used for for confined space, high angle, or technical rescue. SKED© is not an acronym; the word came from fusing two words: "Sled" and "Skid." Over the last several years, as recommendations for spinal protection and utilization of adjunct field hardware for patient application changes, there have been conflicting training and practice regarding optimizing patient packaging utilizing the SKED© system. Specifically, there is disagreement in terms of optimal packaging to ensure no decompensation of respiratory status of the patient objectively, as well as comfort level subjectively solely related to the packaging method utilized. Several training bodies currently employ different practices of packaging including use of an Oregon Spine Splint-II© (OSS-II) system within a SKED©, foam padding, vacuum mattress configuration, or even no additional adjunct at all. The objective of this study is to determine whether adjuncts to the SKED© system impact respiratory physiology, or patient comfort while being dragged over horizontal ground.

DETAILED DESCRIPTION:
This study will be a randomized controlled, non-blinded trial The setting of this study will be an area of level ground, outdoors at a state park. Study enrollment goal is 50 subjects. This was determined by review of statistics from similar studies, available funding and time frame allocated to complete the study. There is not planned interim analysis, and no criteria for ending the study early. Each participant will be packaged using a SKED© system with no assumed spinal injury. Each subject will be packaged with SKED© only; SKED©+OSS-II©; SKED©+Vacuum mattress; SKED©+foam padding. Each patient packaged within their respective systems as one unit will be subject to a 30 meter controlled drag over terrain chosen to mimic a standard dry backcountry extrication drag. Then carried back to the start by a 4 person carry team to simulate a carry out scenario. The same 30 meter ground area will be used for all systems. Built in safety during the drag includes a manually monitored electric winch system with load cells and two safety operators walking alongside the packaged patient. Target movement will be approximately 1.5-2 miles per hour.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Pregnant females
* Incarcerated individuals
* Anyone with difficulty with enclosed or restrictive spaces
* Subjects with a history of lung disease such as Chronic obstructive pulmonary disease (COPD) or asthma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Likert Pain Scale | Minute 1
  Score ranges from 0-10 with a higher score denoting more pain.
Likert Pain Scale | Minute 5
  Score ranges from 0-10 with a higher score denoting more pain.
Borg Dyspnea scale | Minute 1
  Measures difficulty breathing. Score ranges from 0-10 with higher score denoting more breathlessness.
Borg Dyspnea scale | Minute 5
  Measures difficulty breathing. Score ranges from 0-10 with higher score denoting more breathlessness.
Change in End-Tidal Carbon Dioxide (ETCO2) | Between baseline and minute 5
  Change in measurement from baseline.
Change in Pulse Oximetry | Between baseline and minute 5
  Test used to measure the oxygen level (oxygen saturation) of the blood. Oximetry will be compared between interventions and baseline.
Change in Heart Rate | Between baseline and minute 5
  Change in beats per minute from baseline
Change in Respiratory Rate | Between baseline and minute 5.
  Change in breaths per minute from baseline.
Change in Spirometry values for Forced Vital Capacity (FVC) | Between baseline and minute 5
  FVC is the maximum amount of air a person can expel from the lungs after a maximum inhalation. Change in FVC from baseline.
Change in Spirometry values for Forced Expiratory Volume in 6 seconds (FEV6) | Between baseline and minute 5
  FEV6 is the volume of air forcefully exhaled after 6 seconds. Change in FEV6 from baseline.
Change in Spirometry values for Maximal Voluntary Ventilation (MVV) | Between baseline and minute 5
  MVV is a spirometry test that measures the. largest volume that can be moved into and out of the lungs during a 10-15 second interval with voluntary effort. Change in MVV from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Davis, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No